CLINICAL TRIAL: NCT03197116
Title: The Effectiveness of Telephone Reminders by a Layperson on Compliance With Colorectal Cancer Screening: an Open-label, Randomized Controlled Trial
Brief Title: Lay Tel Compliance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Martin Chi Sang Wong, Director, CUHK Jocky Club Bowel Cancer Education Centre, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Lay Tel Compliance
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: CRC Screening; Compliance, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone reminder (Active Comparator): Interactive telephone reminder by a trained layperson with a standard script to remind return to the center for taking fecal tubes for CRC screening
  Interventions: Other: Telephone reminder
- No reminder (Placebo Comparator): No additional reminder will be offered
  Interventions: Other: No other

INTERVENTIONS:
Other: Telephone reminder — Interactive telephone reminder by a trained layperson with a standard script to remind return to the center for taking fecal tubes for CRC screening
  Arms: Telephone reminder
Other: No other — No additional reminder will be offered
  Arms: No reminder

SUMMARY:
This is a randomized controlled study to compare the effectiveness of interactive telephone reminders by a layperson on enhancing compliance with CRC screening by FOBT, when compared with usual care (i.e. no intervention).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the major global health challenges. CRC is currently the third most common cancer in men and the second common in women worldwide, accounting for approximately 10% of all cancers. It leads to 8% of all cancer mortality in the world and it is the fourth most common cause of cancer deaths. There were 4,563 new cases and 3,893 new deaths in Hong Kong in 2012, while 47.4% of the new cases were diagnosed at stage III or above. In the past decades the Asia Pacific countries like China, South Korea, Japan, and Singapore have witnessed a two to three-fold rise in incidence, gradually catching up the figures in Western countries. The direct medical cost for the care of colorectal neoplasia was estimated US$45,115 for stage IV CRC in the initial year of care, bringing a substantial, global public health burden to the healthcare systems.

Randomized controlled studies have shown that CRC screening using Faecal Occult Blood Testing (FOBT) is effective in reducing cancer mortality by 15-33%. FOBT as a quick office-based procedure has the advantages of being non-invasive, inexpensive, acceptable, feasible, patient-friendly and devoid of needs for bowel preparation. A 25% relative risk reduction in CRC mortality was found for those attending at least one round of FOBT screening, according to a systematic review conducted in 2007. Guidelines from the US Preventive Services Task Force, the European Nations, the Asia Pacific Consensus statements and other authorities recommended FOBT as one of the first-line screening modalities, especially in resource-limited regions. Since yearly testing is recommended to maintain programmatic effectiveness, longitudinal adherence is a critical component of FOBT-based screening programs. Our previous study conducted in Hong Kong showed that the rate of compliance with CRC screening was declining since the first year of enrolment.

Nevertheless, it remains unknown whether interventions based on reminder systems could effectively enhance longitudinal compliance with FOBT, especially among those who have already enrolled in a CRC screening programme. Current evidence does not adequately compare whether interactive reminder are superior to usual care (i.e. no reminders).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who joined the bowel cancer screening programme in the CUHK JC Bowel Cancer Education Centre who are expected to follow-up and return to the centre for annual Fecal Occult Blood Test.

Exclusion Criteria:

* (1) had medical conditions rendering them unable to understand telephone; or (2) had no mobile phone were excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
compliance rate of FOBT completion | 6 months
  Rate of completion of FOBT in the year of receiving the interventions/control

SECONDARY OUTCOMES:
compliance rate of FOBT pick up | 6 months
  Rate of return to the centre for taking FOBT tubes in the year of receiving the interventions/control

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No